CLINICAL TRIAL: NCT06145659
Title: Educational-Clinical Linkage to Improve Health Equity for Children With Developmental Delays and Disabilities From Marginalized Communities
Brief Title: School-based Support for Pre-school Aged Children With Developmental Disabilities and Delays
Acronym: PreM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023-1361; R01NR021155 (NIH)
Record Dates: First submitted 2023-11-07; First posted 2023-11-24 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Developmental Delay
Keywords: primary care; implementation; linkage
MeSH Terms: conditions — Learning Disabilities | interventions — Schools, Nursery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linkage Model (Experimental): Preschool and Me intervention
  Interventions: Behavioral: Preschool and Me
- Treatment as Usual (No Intervention): Preschool and Me intervention is not used

INTERVENTIONS:
Behavioral: Preschool and Me — Utilizes patient navigation services and a medical-educational care plan to support linkages between medical and educational systems
  Arms: Linkage Model

SUMMARY:
This proposal aims to test whether a proposed community-clinical linkage (CCL), an educational-medical linkage model, improves access to school-based services and subsequent child, parent, family and health service outcomes and offers a promising strategy to address longstanding racial, ethnic and income health care disparities among families with preschool children with developmental delays and disabilities. The investigators designed an educational-clinical linkage model, Preschool and Me (PreM) which incorporates key components of a CCL. It also utilizes a personalized medical-education care plan with remote lay navigator support to increase access to school-based services.

DETAILED DESCRIPTION:
Participants (n=320) will be randomized to either: 1) 6 months of PreM (intervention group) or 2) a waitlist control arm receiving the intervention after a 6-month delay. All participants will be followed for 12 months with data collection occurring at 4 timepoints (baseline, 3-, 6- and 12-months). There will also be a simultaneously conducted mixed-methods implementation evaluation focusing on implementation outcomes to serve as indicators for implementation success; measures of implementation quality; and intermediate outcomes to understand and address successes and failures in relation to clinical outcomes.

ELIGIBILITY:
Parent-child dyads who meet inclusion criteria will be enrolled.

Child inclusion criteria are:

1. Meets age requirements for early childhood special education (ECSE) services for Illinois (i.e., 3-5 years old);
2. diagnosed with a developmental delay or disability (DD) or determined to be at risk for DD (clinical concerns raised by primary care provider/healthcare provider or by parents at the time of enrollment);
3. is not receiving any ECSE services.

Exclusion Criteria:

if inclusion criteria is met, no other exclusion criteria will be applied.

Parent inclusion criteria are:

1. aged18 years or older;
2. lives in Chicago;
3. speaks English or Spanish;
4. a legal guardian of a child who meets inclusion criteria.

Min Age: 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Percent of children who enroll in a designated early childhood special education (ECSE) program or Chicago Public School | Up to 12 months
  Increased access to early childhood special education (ECSE) as measured by enrollment in designated Chicago Early Learning Education Program or Chicago Public School
Percent of children who receive school-based therapies | Up to 12 months
  Increased access to early childhood special education (ECSE) services as measured by receipt of school-based services
Timeliness of ECSE services | Up to 12 months
  Calculate the time (number of days) from a child's 3rd birthday to 1) date of Individualized Education Plan (IEP) request; 2) date of IEP eligibility meeting; 3) attendance at preschool (first day); and 4) start date of first school-based therapy for those found eligible.
Percent of children who complete each step of IEP process | up to 12 months
  Percent of children who complete each step of IEP process

SECONDARY OUTCOMES:
Child quality of life | Baseline, 12 month follow up
  Child quality of life will be assessed using questionnaires from the Patient Reported Outcomes Measurement Information System (PROMIS). The questionnaires will examine quality of life under the follow domains: well being, relationships, emotional distress, and health. The questionnaires utilize a 5-point likert scale with higher scores reflecting more of the measured construct within the domain.
Child sleep habits | Baseline, 12 month follow up
  Exploratory outcome assessing sleep disturbance using the PROMIS Parent Proxy Sleep Disturbance questionnaire. This 8 question survey of sleep disturbances is scored on a 5-point scale. A higher score indicates poorer sleep hygiene.
Parenting stress | Baseline, 12 month follow up
  Caregiver Strain Short Form consists of 11 items assessing the level of strain caregivers experience in caring for their child consisting of the following factors: objective strain, subjective internalized strain, and subjective externalized strain. Items are rated on a 5-point Likert-type scale that ranges from 1 (not at all) to 5 (very much). Higher scores represent greater strain.
Family Functioning | Baseline, 12 month follow up
  General Functioning 12-item subscale (GF12) of The McMaster Family Assessment Device (FAD); The FAD consists of 7 scales: affective involvement, affective responsiveness, behavioral control, communication, problem solving, roles and general family functioning. Participants are asked to rate how well each statement describes their family on a 4 point scale. Higher scores indicate worse levels of family functioning.
Family-centered care self-assessment tool | Baseline, 12 month follow up
  Family Centered Care Assessment Tool Community Systems of Services and Supports and Community Systems Integration and Care Coordination examines a participants perception of family-centered care received at their healthcare facility; Each item is rated on a 4-point Likert scale (1= never; 4= always) with higher scores indicating a greater perception of family-centered care.
Satisfaction with the Interpersonal Relationship with the Navigator (PSN-I) | Up to 6 months
  Satisfaction with the Interpersonal Relationship with the Navigator (PSN-I) is a 9 item questionnaire that examines participants perception of their PreM navigator; Each item is rated on a 5-point Likert scale with a higher score indicating a higher satisfaction with their interpersonal relationship with the patient navigator.
Acceptability of Intervention Measure | Up to 6 months
  Acceptability of Intervention Measure examines participants acceptability of PreM; Each item is rated on a 5-point Likert scale with a higher score indicating a greater acceptability
Adoption | up to 6 months
  Ratio of number of Primary Care Providers (PCPs) who referred to Preschool and Me (PreM) to total number of PCPs
Intervention Appropriateness Measure (IAM) | up to 6 months
  Intervention Appropriate Measure examines perception of the appropriateness of PreM; Each item is rated on a 5-point Likert scale with a higher score indicating a greater perception of appropriateness
Penetration | up to 6 months
  Ratio of number of caregivers contacted by Patient Navigator (PN) to number of caregivers referred
Feasibility of Intervention Measure | up to 6 months
  Feasibility of Intervention Measure examines perception of the feasibility of PreM; Each item is rated on a 5-point Likert scale with a higher score indicating a greater perception of feasibility
Fidelity | up to 6 months
  Per family ratio of number of PN activities conducted to number of activities that should be conducted according to protocol/job aid
Cost | up to 6 months
  Time estimates of training and supervision; Per family time estimates associated with PN activities
Parental Quality of Life | Baseline and 12 months
  Parent Quality of Life will be assessed using PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 6a which examines satisfaction with performing one's social roles and activities. Higher scores reflect more of the measured construct (i.e., ability to participate in social roles and activities).

OTHER OUTCOMES:
Positive Protective Factors (Resilience, Social Connections, Concrete Support in Time of Need) | 6, 12 months
  Parent Assessment of Protective Factors is a measure to assess participants' self-reported beliefs, feelings, and behaviors in the areas of Resilience, Social Connections, Concrete Support in Time of Need. Items are scored on a 5 point Likert scales with higher scores indicating a higher perceived strength level.
Parent Patient Activation Measure Parent Patient Activation Measure Parent Patient Activation Measure | 6, 12 months
  Parent Patient Activation Measure assesses perceived knowledge, skills, and confidence in managing child's care. Items are scored using a 4-point Likert scale (1 = disagree strongly; 4 = agree strongly). Higher scores correspond to higher activation.

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Shah, MD, MPH, Principal Investigator — University of Illinois at Chicago
Locations (1):
- UI Health, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) with all potentially identifying information removed will be shared. IPD from a study publication will be shared at the time of publication. Study data will be shared approximately 12 months following the end of data collection but within the funded award period. IPD to be shared includes individual level survey and questionnaire data, coded interview data, and coded data abstracted from the child's medical record, Individualized Education Plan (if applicable), domain specific Early Childhood Special Education therapies, educational placement and supports.
Supporting Information: Study Protocol, ICF
Time Frame: IPD from a study publication will be shared at the time of publication. Study data will be shared approximately 12 months following the end of data collection but within the funded award period.
Access Criteria: The final study data and documentation will be made available to researchers through the Interuniversity Consortium for Political and Social Research (ICPSR) repository services. Access to data underlying publications will vary based on the publication and information on access will be available either in the publication or made available by the study PI.